CLINICAL TRIAL: NCT01092754
Title: An Open-Label, Multicenter, Phase 4 Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Optimark(R) in Pediatric Patients (2-11 & 12-18 Yrs) Referred for Contrast-Enhanced MRI
Brief Title: Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Optimark (Gadoversetamide) in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Eddie Darton, Jr., M.D./Director, Global Drug Safety & PVG, Mallinckrodt Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1177-01-597
Record Dates: First submitted 2010-03-15; First posted 2010-03-25 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Pathological Processes
Keywords: brain, spine, liver, MRI, Pediatric
MeSH Terms: conditions — Pathologic Processes | interventions — gadoversetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Other (Other)
  Interventions: Procedure: MRI; Drug: Gadoversetamide
- B: Other (Other)
  Interventions: Procedure: MRI; Drug: Gadoversetamide

INTERVENTIONS:
Procedure: MRI — contrast enhanced MRI
  Other Names: gadoversetamide
  Arms: A: Other
Procedure: MRI — contrast enhanced MRI
  Other Names: gadoversetamide
  Arms: B: Other
Drug: Gadoversetamide — Subjects will receive a single dose of Optimark(0.1 mmol/kg)as a bolus thru a peripheral IV line at 1-2 mL/sec followed by a saline flush during their medically necessary MRI .

SUMMARY:
The objective of this study is to characterize the safety, efficacy and pharmacokinetic profiles of Optimark at the standard clinical dose of 0.1 mmol/kg in the pediatric patient population.

DETAILED DESCRIPTION:
Pediatric patients referred for magnetic resonance imaging (MRI) of the liver or central nervous system (CNS) will be stratified by age to one of two groups (2 through 11 and 12 through 18 years of age).

ELIGIBILITY:
Inclusion Criteria:

* 2 thru 18 years of age
* referred for MRI of the liver or CNS
* if female and of child-bearing potential, must have negative pregnancy test within 24 hours of study drug administration
* if applicable, agree to use medically accepted method of contraception throughout the study
* if necessary, patients entering the PK subgroup must be willing to be housed within the investigational facility for a minimum of 24 hours following drug administration
* understand the requirements of the study and provide written consent to participate, agree to abide by the study requirements

Exclusion Criteria:

* previously entered into this study or a previous study using Optimark
* received investigational drug within 30 days of admission into this study or plan to participate in a clinical study prior to the end of this study's monitoring period. (patients on a research protocol using an approved drug ar acceptable)
* medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance and all prescribed follow up
* known or suspected abnormal renal function for age or requiring dialysis during the study period
* pregnant or breastfeeding
* scheduled to undergo any contrast-enhanced examination within 7 days prior to baseline examination or during the course of this study period
* condition that is a contraindication to MRI (i.e., cardiac pacemaker, epicardial pacemaker leads, cochlear implants, ferromagnetic aneurysm clip, ferromagnetic halo device, or other condition that would preclude patient proximity to a strong external magnetic field)
* experienced a previous hypersensitivity reaction to a gadolinium-based contrast agent
* recent history of hemolytic anemia, sickle cell anemia, or other hemoglobinopathy
* undergone a surgical procedure within one week prior to study admission or are planned to undergo a surgical procedure during study participation (central line placement is acceptable)
* history of significant claustrophobia
* weighs less than 25 lbs (11 kgs)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2002-05; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Assess efficacy by analyzing the clinical diagnosis, degree of confidence in diagnosis and level of conspicuity of lesions. | Immediately before and immediately after Optimark dosing
  Optimark is an MRI contrast. Efficacy measurements will be determined from images obtained without contrast (immediately before) and with contrast (immediately after).

SECONDARY OUTCOMES:
Assess the safety of Optimark by analyzing adverse events and changes in vital signs, electrocardiograms (ECGs), physical exams, and clinical laboratory results. | through 24 hours post dose
Assess the blood and urine PK levels of Optimark | through 10 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Darton, MD, Study Chair — Mallinckrodt
Locations (12):
- United States (12):
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Childrens Hospital and Health Center, San Diego, California
  - Miami Children's Hospital, Miami, Florida
  - Children's Mercy Hospitals and clinics, Kansas City, Kansas
  - Louisiana State University Sciences Center- Shreveport, Shreveport, Louisiana
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Cardinal Glennon Childrens Hospital, St Louis, Missouri
  - St. Louis Childrens Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Childrens Hospital, Houston, Texas